CLINICAL TRIAL: NCT04436172
Title: Spinal Anesthesia Facilitated Sexual Intercourse As A Treatment Option For Vaginismus And Its Effect On Female Sexual Dysfunction As Assessed By Female Sexual Functioning Index (Fsfi) - A Pre-Post Intervention Design Study
Brief Title: Spinal Anesthesia Facilitated Sexual Intercourse As A Treatment Option For Vaginismus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karachi Medical and Dental College (Other)
Collaborators: Aziz Medical Center (Network)
Responsible Party: Principal Investigator, samia husain, clinical investigator, Karachi Medical and Dental College
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KarchiMDC
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Vaginismus
MeSH Terms: conditions — Vaginismus | interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre intervention (No Intervention): Before intervention
- post intervention (Experimental): Received soinal anesthesia
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — The spinal anesthesia was given by a trained anesthetist in an equipped room, after all aseptic measures. A 20 gauge intravenous cannula was inserted for maintaining a peripheral line and 0.9% normal saline was used for loading the patient. The pulse and blood pressure were monitored non-invasively. The median approach was utilized and intrathecal space was accessed via 25 gauge Quiincke bevel(Becton Dickinson/Pakistan ) through L4-L5. A block was performed by using 5 mg hyperbaric bupivacaine (Abocain 0.5%/Abbot) after ensuring swirling. Block height was monitored via pinprick test after every three minutes, for 20 minutes until there was no progression. The couple was left alone. The couples received prior training and were explained precautions.
  Arms: post intervention

SUMMARY:
Painful sex continues to be a relationship issue and can lead to marital dys-harmony. Other consequences include infertility, low self-esteem, depression and anxiety.Our study shows that spinal anesthesia is an effective last resort management option in women with vaginismus. As a one-off treatment spinal anesthesia provides hope for such couples and brings about a positive change in their relationships.

ELIGIBILITY:
Inclusion Criteria:

* Virgin married women with non-consummation of marriage for more than two years due to vaginismus

Exclusion Criteria:

* partners reported erectile dysfunction
* who had vulvar skin conditions (e.g. lichen sclerosus)
* vulvovaginal and urinary tract infections
* endometriosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
successful sexual intercourse | 1 year
  whether couple was able to have sexual intercourse after treatment
improvement in Female sexual functioning index | 1 year
  Female sexual function index (FSFI) questionnaire consists of 19 questions that assess 6 domains to assess sexual feelings and responses during the past 4 weeks.

SECONDARY OUTCOMES:
depression and relationship satisfaction | 1 year
  Depression was assessed by Zung's score. Zung's Self-Rating Depression Scale is a twenty item likert scale with raw score that ranges from 20 to 80. There are 20 items on the scale that rate the four common characteristics of depression: the pervasive effect, the physiological equivalents, other disturbances, and psychomotor activities.
  Relationaship assessment was assesed by relationship assessment score.The Relationship Assessment Scale (RAS) is a brief measure of global relationship satisfaction.

IPD SHARING:
Plan to Share IPD: No